CLINICAL TRIAL: NCT05506943
Title: A Phase 2/3 Randomized, Controlled Study of CTX-009 in Combination With Paclitaxel Versus Paclitaxel Alone in Adult Patients With Unresectable Advanced, Metastatic or Recurrent Biliary Tract Cancers Who Have Received One Prior Systemic Chemotherapy Regimen
Brief Title: A Study of CTX-009 in Combination With Paclitaxel in Adult Patients With Unresectable Advanced, Metastatic or Recurrent Biliary Tract Cancers (COMPANION-002)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Compass Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTX-009-002
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma; Gall Bladder Cancer; Ampullary Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded independent review committee will be used to assess the primary study endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTX-009 plus Paclitaxel (Experimental)
  Interventions: Drug: CTX-009; Drug: Paclitaxel
- Paclitaxel (Active Comparator): Patients randomized to receive paclitaxel only have the option to crossover to the CTX-009 plus paclitaxel arm after documented disease progression per RECIST v1.1.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: CTX-009 — IV infusion on day 1 and 14 of every 28 day cycle
  Arms: CTX-009 plus Paclitaxel
Drug: Paclitaxel — IV infusion on day 1, 8, and 15 of every 28 day cycle

SUMMARY:
This is a multi-center, open-label, randomized, phase 2/3 trial of the bispecific antibody CTX-009 plus paclitaxel versus paclitaxel in patients with previously treated, unresectable advanced or metastatic biliary tract cancers.

ELIGIBILITY:
INCLUSION CRITERIA

1. 18 years of age or older
2. Histologically or cytologically confirmed unresectable advanced, metastatic, or recurrent biliary tract cancers (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, gallbladder cancer, and ampullary carcinoma)
3. Patients must have radiologically documented progression after a prior gemcitabine and platinum containing chemotherapy regimen as first line therapy for locally advanced unresectable or metastatic disease.

   1. Patients who received perioperative treatment (adjuvant and neoadjuvant) may be eligible, as determined by the Sponsor Medical Monitor.
   2. Patients whose first line regimen was modified due to toxicity before disease progression, may be eligible, as determined by the Sponsor Medical Monitor.
4. At least one lesion measurable as defined by RECIST v1.1
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
6. Predicted life expectancy of at least 12 weeks
7. No evidence of ongoing infection and adequate biliary excretion or patients whose adequate biliary excretion can be confirmed with the following procedures:

   1. Patients who underwent endoscopic retrograde biliary drainage (ERBD) at least 1 week before the investigational drug treatment
   2. Patients with endobiliary stents are eligible, provided there is no evidence of obstruction
   3. Patients free of any signs of active or suspected uncontrolled infection after a drainage procedure
   4. Patients free of any risk of hemorrhage and with incision completely healed
8. Adequate bone marrow, hepatic, and renal function within 14 days of randomization as described below. (Patient must be free of G-CSF treatment and blood transfusion within 14 days prior to the lab test):

   1. Absolute neutrophil count (ANC) ≥ 1,500/mm3
   2. Hemoglobin ≥ 9.0 g/dL
   3. Platelet count ≥ 100,000/mm3
   4. Total bilirubin ≤ 1.5 X ULN
   5. AST/ALT ≤ 3.0 X ULN (≤5 X ULN in case of hepatic metastasis)
   6. Estimated creatinine clearance ≥ 30 mL/min based on Cockcroft-Gault
   7. Urine protein ≤ 1+ by Dipstick (Only when urinalysis shows a protein dipstick result of > 1 positive (+), the total protein volume (<1.0 g/24hr) can be confirmed with a 24-hour urine test.)
   8. Serum amylase and lipase level ≤ 3X ULN
   9. Serum Albumin ≥ 3.0 g/dL
9. Female patients who are women of childbearing potential (WCBP) must have a negative pregnancy test (serum-hCG or urine-hCG performed at the Investigator's discretion) within 14 days of randomization
10. Female patients must be surgically sterile (or have a monogamous partner who is surgically sterile) or be at least 2 years postmenopausal or commit to use 2 acceptable forms of birth control (defined as the use of an intrauterine device (IUD), a barrier method with spermicide, condoms, or any form of hormonal contraceptives) or abstinence for the duration of the study and for 6 months following the last dose of study treatment. Male patients must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for 6 months following the last dose of study treatment.
11. Signed and dated Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved Informed Consent Form (ICF) before any protocol-directed screening procedures are performed

EXCLUSION CRITERIA

1. Patients who are eligible to be treated with a molecularly targeted therapy on a labelled regimen after receiving first-line chemotherapy. Patients who received a molecularly targeted therapy as part of their first line treatment may be eligible, as determined by the Sponsor Medical Monitor.
2. From the time point of screening,

   1. Less than 4 weeks have elapsed since patients had a surgery or major procedure
   2. Less than 2 weeks have elapsed from the last treatment date since patients had any radiation therapy
3. Patients with percutaneous transhepatic biliary drains (PTBD)
4. Prior to the initial treatment of study drug,

   1. Less than 2 weeks have elapsed since patients had chemotherapy or hormone therapy
   2. Less than 2 weeks have elapsed since patients had anticancer immunotherapy or investigational drug treatment
   3. Less than 4 weeks since cryotherapy, radiofrequency ablation, anhydrous alcohol therapy, or photodynamic therapy, including TACE and TARE
5. A history of the following cardiovascular diseases (please, consult the Sponsor Medical Monitor for a case by case evaluation):

   1. Congestive heart failure (CHF) that corresponds to Class II or a higher class under New York Heart Association (NYHA) classification, or less than 50% of left ventricular ejection fraction (LVEF)
   2. Uncontrolled hypertension (SBP/DBP >140/90 mmHg) (e.g., patient with SBP/DBP >140/90 mmHg despite the best care including optimizing the anti-hypertensive medication regimen)
   3. Patients with any history of hypertensive crisis or pre-existing hypertensive encephalopathy
   4. Pulmonary hypertension
   5. Myocardial infarction
   6. Uncontrolled arrhythmia
   7. Unstable angina
   8. Patients with any significant vascular diseases (e.g., aortic aneurysm requiring surgery or recent peripheral artery thrombosis) within 6 months prior to the initial treatment of the investigational product
6. History of hypersensitivity reactions to any components of the investigational product or other drugs of the same class (humanized/human monoclonal antibody drugs) or paclitaxel
7. Patients with contraindications to paclitaxel therapy
8. Patients with persistent, clinically significant toxicities (excluding hair loss) from previous anticancer treatment that corresponds to Grade 2 or a higher grade under NCI-CTCAE v5.0
9. Symptomatic or uncontrolled central nervous system (CNS) metastasis (However, patients with asymptomatic CNS metastasis that have been treated with either surgery or radiation can participate provided that systemic corticosteroid treatment was discontinued at least 4 weeks prior to screening and that the patient is radiologically and neurologically stable or improving)
10. A history of the following hemorrhage-related or gastroenterological disease:

    1. Active hemorrhage, hemorrhagic diathesis, coagulopathy or tumor in great arteries
    2. History of clinically significant gastroenterological disease, such as peptic ulcer, GI bleeding, GI or non-GI fistula, perforation, abdominal abscess, clinical symptoms, and signs of GI obstruction, need for parenteral hydration or nutrition, or inflammatory bowel disease (IBD)
11. Current or recent (within 10 days prior to study treatment) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose will be excluded.

    a. Prophylactic (i.e., for the patency of venous access devices) use of low molecular weight heparin (i.e., enoxaparin 40 mg/day) is allowed if patient has INR < 2 or aPTT </=2x ULN within 14 days of study treatment
12. Patients with current or recent (within 10 days of study treatment) use of aspirin (>81 mg/day), or other nonsteroidal anti-inflammatory drugs (NSAIDs), or other antiplatelets (i.e., dipyramidole, ticlopidine, clopidogrel, and cilostazol) will be excluded.
13. Severe infection requiring ongoing systemic antibiotics, antivirus drugs, etc., or other uncontrolled acute active infectious diseases
14. Patients with evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with positive HBsAg and/or detectable HBV DNA are eligible only if adequately controlled on antiviral therapy according to institutional standards and liver function eligibility criteria are also met. HCV patients showing sustained viral response or patients with immunity to HBV infection may enroll.
15. Patients with other severe diseases or uncontrolled illnesses that warrant the exclusion from the study (permitted only if medically controlled) including but not limited to:

    1. Pre-existing hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 28 days prior to screening
    2. Major, unhealed injury, active ulcer, or untreated fracture
    3. Pre-existing conditions of cerebrovascular incident (ischemic or hemorrhagic stroke), transient ischemic attack or subarachnoid hemorrhage within 6 months prior to screening.
    4. Moderate to severe ascites and/or pleural effusion. However, enrollment is permitted for patients with ascitic fluid as long as paracentesis is not required to improve the condition.
    5. Interstitial lung disease or pulmonary fibrosis
16. Patients expected to require anticancer treatment other than the investigational product during the clinical study
17. Pregnant or lactating patients, or patients planning to become pregnant during the clinical study
18. A history of primary malignancy other than BTC will be excluded, except for malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%). Prior malignancy history will be evaluated on a case-by-case basis by the Sponsor Medical Monitor.
19. Clinically significant abnormal ECG findings or history determined as clinically significant by the Investigator
20. QT interval (Fridericia's formula) (QTcF) interval > 450msec at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response | From randomization to treatment discontinuation for any reason, average 6 months
  Percentage of patients whose Best Overall Response (BOR) is assessed as Complete Response (CR) or Partial Response (PR) as assessed by RECIST 1.1

SECONDARY OUTCOMES:
Progression Free Survival | From randomization to first documented objective PD or death if PD does not occur, average 6 months
  Time from randomization until the date of objective PD (as assessed by RECIST 1.1) or the date of death (by any cause in the absence of disease progression)
Duration of Response | From first confirmed CR or PR to confirmed PD, average 6 months
  The time between the date of the radiological evaluation that first confirmed CR or PR and the date of the radiation evaluation that first confirmed Progressive Disease (PD)
Overall Survival | From randomization to death from any cause, average 12 months
  Time from randomization until the date of death by any cause. Patients who are still alive at the time of the analysis, or who have become lost to follow-up or withdrawn consent will be censored at their last date known to be alive
Disease Control Rate | From randomization to treatment discontinuation for any reason, average 6 months
  Percentage of patients whose BOR is assessed as CR, PR, or Stable Disease (SD)
Safety Profile of CTX-009 in Combination with Paclitaxel | From randomization to 60 days after the last dose of study treatment, average 7 months
  Incidence of Treatment Emergent Adverse Events (TEAEs) and changes in clinical abnormalities for all randomized patients who received at least one dose of study treatment (either CTX-009 or paclitaxel)
Patient Reported Quality of Life | From randomization to treatment discontinuation for any reason, average 6 months
  Assessed approximately every 2 months from patient reported data using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (QLQ)-C30 and BIL21
Exposure Response by Pharmacokinetic (PK) Sampling | From C1D1 to treatment discontinuation for any reason, average of 6 months
  Serum concentrations of CTX-009 at specified timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Minori Rosales, MD, PHD, Study Director — Compass Therapeutics
Locations (34):
- United States (34):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Medicine Cancer Center, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - The University of New Mexico, Albuquerque, New Mexico
  - Memorial Medical Center, Las Cruces, New Mexico
  - Roswell Park, Buffalo, New York
  - Columbia University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Dension, Denison, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Mason Franciscan Health, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azad N, Hu Z, Sahin I, Iyer R, Aranha O, Hochster H, Pathak P, Paulson AS, Kalyan A, Liao CY, Tran N, Kelley RK, Heestand G, Cosgrove D, El-Khoueiry A, Borad M, Gabrail NY, Majeed U, Du L, Kamath S, Shumway N, Shroff R, Goyal L, Rosales M, Javle M. COMPANION-002 A clinical trial of investigational drug CTX-009 plus paclitaxel vs paclitaxel in second line advanced BTC. Future Oncol. 2024;20(30):2241-2248. doi: 10.1080/14796694.2024.2351351. Epub 2024 Jun 4. PMID 38861293